CLINICAL TRIAL: NCT05421429
Title: An Open, Multicenter, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous (SC) Doses of KN057 in Subjects with Hemophilia a or B, with or Without Inhibitors
Brief Title: KN057 Multiple Dose Study in Moderately Severe to Severe Hemophilia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: KN057-A-201
Record Dates: First submitted 2022-06-09; First posted 2022-06-16 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- KN057 (Cohort 1：HA/HB) (Experimental): Injection, once a week
  Interventions: Biological: KN057 doseⅠ
- KN057 (Cohort 2：HA/HB) (Experimental): Injection, once a week
  Interventions: Biological: KN057 dose Ⅱ
- KN057 (Cohort 3：HA/HB) (Experimental): Injection, once a week
  Interventions: Biological: KN057 dose Ⅱ
- KN057 (Cohort 4：HAW/HBW) (Experimental): Injection, once a week
  Interventions: Biological: KN057 dose Ⅲ

INTERVENTIONS:
Biological: KN057 doseⅠ — KN057 subcutaneous (SC) injection
  Arms: KN057 (Cohort 1：HA/HB)
Biological: KN057 dose Ⅱ — KN057 SC injection
  Arms: KN057 (Cohort 2：HA/HB); KN057 (Cohort 3：HA/HB)
Biological: KN057 dose Ⅲ — KN057 SC injection
  Arms: KN057 (Cohort 4：HAW/HBW)

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of multiple subcutaneous doses of KN057 in subjects with hemophilia A or B, with or without inhibitors to Factor VIII (FVIII) or Factor IX (FIX). 24 adult participants 18 to 70 years of age with moderately severe to severe hemophilia A or hemophilia B (defined as FVIII or FIX activity ≤2%, respectively) with or without inhibitors (including 18 HA/HB patients without inhibitors and 6 HA/HB patients with inhibitors) are expected to be enrolled in this study during which they will receive prophylaxis treatment (defined as treatment by SC injection once weekly of KN057).

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18-70 years old (including threshold), weight≥40kg;
2. Moderately severe to severe hemophilia A or B (Factor VIII or Factor IX activity ≤2%)
3. Participants who are enrolled into the Non-Inhibitor Cohort must meet the following criteria:

   ①negtive results of of inhibitors to Factor VIII (FVIII) or Factor IX (FIX) in screening period.

   ②with ≥6 acute bleeding episodes (spontaneous or traumatic, not including episodes of bleeding during surgery) that required treatment within 6 months before screening and willing to continue to receive on-demand treatment during the study.

   ③using coagulation factor replacement therapy for more than 50 exposure days before screening.
4. Participants who are enrolled into the Inhibitor Cohort must meet the following criteria:

   ①positive results of inhibitors to Factor VIII (FVIII) or Factor IX (FIX) in screening period.

   ②with ≥6 acute bleeding episodes (spontaneous or traumatic, not including episodes of bleeding during surgery) that required treatment within 6 months before screening and willing to continue to receive on-demand treatment during the study.
5. Be willing to undergo a washout period of the original treatment regimen before the administration of KN057: at least 48 hours for recombinant activated coagulation factor Ⅶ (rFⅦa); at least 72 hours for FⅧ and prothrombin complex (PCC); at least 96 hours for FⅨ; For other drugs or investigational products with a long half-life, such as Emicizumab, at least five half-lives should have passed prior to dosing.
6. Be willing to comply with the relevant management regulations of the clinical trial unit, and follow study procedures.

Exclusion Criteria:

1. Patients with serious or poorly controlled chronic diseases or obvious systemic diseases, such as cardiovascular system, respiratory system, endocrine and metabolic system, urinary system, digestive system, autoimmune diseases, nervous system diseases or psychiatric diseases, bacterial or viral infections, etc.; past or current lipid-lowering treatment for hypertriglyceridemia.
2. Inherited or acquired bleeding disorder other than hemophilia A or B.
3. Have symptoms or signs related to thromboembolic disease or are receiving thrombolytic/anti-thrombolytic therapy; A history of coronary atherosclerotic diseases, arterial or venous thrombosis, and ischemic diseases of important organs.
4. Conditions that may increase risk of thrombosis: including reduced activity of antithrombin III, protein S or protein C;
5. Must use PCC to treat acute bleeding episodes, and can't be treated with rFVIIa.
6. Ongoing or planned use of immune tolerance induction.
7. Regular use of immunomodulatory therapy, such as regular infusion of immunoglobulin or regular use of hormones.
8. Allergy situation: Allergic to test drugs/similar drugs or excipients; With a history of multiple allergies (two or more); A history of specific reactions, such as sensitivity to heparin or heparin induced thrombocytopenia.
9. Abnormal hematologic parameters: Platelet count≤100×10^9/L; Hemoglobin < 100g/L; Fibrinogen level < LLN; Prothrombin time > 1.5 times ULN;
10. Abnormal renal or hepatic function: Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 times ULN; Lactate dehydrogenase (LDH) > 1.5 times ULN; Total bilirubin (TB) > 1.5 times ULN; Serum creatinine (Cr) and triglyceride > ULN; Albumin < 0.8 times LLN;
11. Chronic active hepatitis B/C (HBV-DNA or HCV-RNA quantitative test indicates viral activity); Human immunodeficiency virus (HIV) antibody positive; Syphilis antibody positive; Previous antiviral treatment within 1 month, or a plan for antiviral treatment within 28 weeks of initial administration.
12. Had major surgery, as judged by the investigator, within 3 months prior to the study or have elective surgery planned within 28 weeks of initial administration.
13. Need to use anti-fibrinolytic drugs or drugs affecting platelet function 5 days before administration or 28 weeks after initial administration, including Traditional Chinese medicine/proprietary Chinese medicine, such as aspirin and other non-steroidal anti-inflammatory drugs, Angelica, astragalus, etc., or proprietary Chinese medicine containing the above ingredients.
14. Participated in clinical trials related to coagulation factors within 1 month; Participated in any other drug clinical trials within 3 months.
15. Vaccination within 1 month, or within 28 weeks after initial administration, including inactivated vaccines, live attenuated vaccines, recombinant protein vaccines, recombinant adenovirus vaccines, RNA vaccines, DNA vaccines, etc.;
16. Subjects with fertile partners are not willing to use effective contraception during the study period and for 3 months after the last dosing; Effective contraceptive methods include: vasectomy, adhere to the scientific use of male condoms, etc.
17. Other factors that the investigator considers unacceptable for participation in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events(TEAEs) | Day 1 up to Day 85
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. A serious adverse event (SAE) is any untoward medical occurrence at any dose that resulted in death; life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and non-serious AEs. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment.
Withdrawals due to TEAEs | Day 1 up to Day 85
  An AE is any untoward medical occurrence in a clinical investigation participant administered a product and the event does not need to have a causal relationship with the treatment. TEAEs are AEs occurred following the start of treatment or AEs increasing in severity during treatment.
Number of Participants With Abnormal Laboratory Findings-Hematology | Day 1 up to Day 85
  White blood cells, red blood cells; the count of lymphocyte, neutrophils, monocytes, eosinophils, basophils; the percentage of lymphocyte, neutrophils, monocytes, eosinophils, basophils; hemoglobin, red blood cell pressure, platelet count
Number of Participants With Abnormal Laboratory Findings-Urinalysis | Day 1 up to Day 85
  blood, urobilirubin, urobiliogen, ketone body, protein, nitrite, red blood cell (qualitative and/or quantitative), white blood cell (qualitative and/or quantitative), pH, urinary glucose.
Number of Participants With Abnormal Laboratory Findings-Blood biochemistry | Day 1 up to Day 85
  Total bilirubin and indirect bilirubin, direct bilirubin, alanine aminotransferase, aspertate aminotransferase, GGTP (gamma glutamyl transpeptidase), alkaline phosphatase, total protein, albumin, globulin, albumin-globulin ratio, urea, creatinine, uric acid, glucose, total cholesterol, triglyceride, low density lipoprotein cholesterol (ldl-c), high-density lipoprotein cholesterol (hdl-c), lactate dehydrogenase, creatine kinase, chlorine, calcium, sodium, potassium, C reactive protein
Number of Participants With Abnormal Laboratory Findings-Coagulation tests | Day 1 up to Day 85
  Prothrombin time (PT), International Standardized ratio (INR), Activated partial thrombin time (APTT), thrombin time (TT), fibrinogen (FBG/FIB), D-dimer (D-DI), fibrinogen degradation product (FDP), antithrombin - ⅲ (AT- ⅲ)
Number of Participants With Clinically Significant Changes in Vital Signs Data | Day 1 up to Day 85
  Vital signs：blood pressure (systolic blood pressure, diastolic blood pressure), respiration, temperature, pulse；
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) | Day 1 up to Day 85
  ECG: HR; RR; PR; QRS; QT; QTc
Number of Participants With Clinically Significant Changes in Physical Examination Findings | Day 1 up to Day 85
  Physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Clinical significance was judged by the investigator.
Number of Participants With Injection Site Reactions | Day 1 up to Day 85
  Injection site reactions may include, but are not limited to: erythema, sclerosis, ecchymosis, pain, and itching.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of KN057 | Day 1 up to Day 8
Time to Reach Maximum Plasma Concentration (Tmax) of KN057 | Day 1 up to Day 8
Area Under the Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of KN057 | Day 1 up to Day 8
Cmax,ss: Maximum observed KN057 concentration at steady-state | Day 36 up to Day 43
Time to Reach Maximum Plasma Concentration at steady-state (Tmax,ss) of KN057 | Day 36 up to Day 43
Area Under the Serum Concentration-time Curve Over the Dosing Interval Tau (AUCtau) of KN057 | Day 36 up to Day 43
Apparent Clearance (CL/F) of KN057 | Day 36 up to Day 43
Lowest Concentration Observed During the Dosing Interval (Cmin) of KN057 | Day 36 up to Day 43
Pharmacodynamics index: Changes of TFPI from baseline; | Day 1 up to Day 169
  Tissue factor (TF) pathway inhibitor (TFPI) is an anticoagulant protein that inhibits early phases of the procoagulant response. TFPI: Total TFPI, Free TFPI
Pharmacodynamics index: Changes of Prothrombin fragment 1+2 (PF1+2) from baseline; | Day 1 up to Day 169
  Prothrombin fragment 1+2 (F1+2) is the amino terminus fragment of the prothrombin molecule.
Pharmacodynamics index: Thrombin Generation (TGA); | Day 1 up to Day 169
  Lag Time; Peak Thrombin; Endogenous Thrombin Potential;
Number of Participants Who Tested Positive for Anti-KN057 Antibody (ADA) | Day 1 up to Day 169
  Human plasma ADA samples were analyzed for the detection of anti KN057 antibodies.
Number of Participants Who Tested Positive for Neutralizing Antibody (NAb) | Day 1 up to Day 169
  Human plasma NAb samples were analyzed for the presence or absence of NAb to KN057.
Annualized Bleeding Rate | Day 1 up to Day 169
  ABR = number of bleeds requiring treatments/ (days on treatment period / 365.25)

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Doctor, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences; Shujie Wang, Doctor, Principal Investigator — Peking Union Medical College Hospital; Hu Zhou, Doctor, Principal Investigator — Henan Cancer Hospital（The Affiliated Cancer Hospital Of ZhengZhou University); Ziqiang Yu, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University; Changcheng Zheng, Doctor, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital); Jing Sun, Doctor, Principal Investigator — Nanfang Hospital, Southern Medical University; Xielan Zhao, Doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - stitute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided